CLINICAL TRIAL: NCT07078409
Title: Clinician Nudge to Referral of Adnexal Masses to Gynecologic Oncology
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Anna Jo Bodurtha Smith, MD, MPH, MSc, Assistant Professor, Gynecologic Oncology, Perelman School of Medicine, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 858390; HT9425-25-1-0243 (Other Grant/Funding Number: DoD)
Record Dates: First submitted 2025-06-25; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer
Keywords: nudge
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nudge (Experimental): When the clinician who ordered the imaging that led to randomization receives the test results, a pre-checked referral order to gynecologic oncology for surgical evaluation will appear in the EHR alongside a brief educational explanation. This will constitute the opt-out default referral order (Figure 3). Clinicians will have the option to unclick the referral to opt out and will be asked to indicate the reason from a pre-populated list of choices; if they do not opt out, the referral to gynecologic oncology will proceed. Imaging findings and referral will be communicated to the patient in keeping with the clinician's usual practice. In keeping with routine practice, referred patients will be contacted by gynecologic oncology's new patient coordinators within 72 hours and offered an appointment within 2 weeks at their preferred location.
  Interventions: Behavioral: Nudge
- Control (No Intervention): Clinicians will receive imaging reports per usual practice (i.e., imaging reports that include O-RADS score with recommendation for gynecologic oncology referral in the report) and can place referral through the usual EHR-based ordering system. If referred, patients will be contacted and scheduled as described above.

INTERVENTIONS:
Behavioral: Nudge — When the clinician who ordered the imaging that led to randomization receives the test results, a pre-checked referral order to gynecologic oncology for surgical evaluation will appear in the EHR alongside a brief educational explanation. This will constitute the opt-out default referral order (Figure 3). Clinicians will have the option to unclick the referral to opt out and will be asked to indicate the reason from a pre-populated list of choices; if they do not opt out, the referral to gynecologic oncology will proceed. Imaging findings and referral will be communicated to the patient in keeping with the clinician's usual practice. In keeping with routine practice, referred patients will be contacted by gynecologic oncology's new patient coordinators within 72 hours and offered an appointment within 2 weeks at their preferred location.
  Arms: Nudge

SUMMARY:
The goal of this study is to test the effectiveness of clinician nudges on referrals to gynecologic oncology in patients with suspected ovarian cancer.

The primary outcome will be whether or not patients were referred to gynecologic oncology within 14 days of their abnormal imaging results. Secondary and exploratory outcomes are whether the gynecologic visit occurred within 60 days of abnormal imaging and the time from abnormal imaging results to gynecologic oncology visit.

ELIGIBILITY:
Inclusion Criteria:

* Eligible clinicians include physicians, physician assistants, and nurse practitioners with eligible patient encounters at sites included in the trial during the study.
* Eligible patient encounters are defined as an emergency room visit, inpatient hospitalization, or outpatient visit during the study period where the patient had associated imaging with suspected ovarian cancer (O-RADS 4 or 5 lesion), identified with the EHR-based tool described above.

Exclusion Criteria:

* Known diagnosis of ovarian cancer.
* Imaging ordered by gynecologic oncologist.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-07-07 (Estimated); Study Completion 2027-07-07 (Estimated)

PRIMARY OUTCOMES:
Referral Rate | Up to one year
  Binary indicator of whether the patient was referred to gynecologic oncology within 14 days of abnormal imaging results.

SECONDARY OUTCOMES:
Gynecologic Oncology Visit | Up to one year
  Whether or not the gynecologic oncology visit occurred within 60 days of abnormal imaging.
Time from imaging to visit | Up to one year
  Time from abnormal imaging results to gynecologic oncology visit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share data arising from the proposed project to the extent that it is permissible and consistent with the prevailing data use agreements and controlling IRBs. Data sharing will occur in a timely fashion.
  Following acceptance for publication of the main findings from the final data set, we will provide for the timely release and sharing of the de-identified data from the cohort study and the qualitative interviews. These data sets will be provided upon written request to all interested investigators. Upon acceptance for publication of the main study findings, we will also share upon written request with interested investigators the code used in analyzing data.
Supporting Information: Study Protocol, SAP
Access Criteria: Beginning 1 year after publication with no end date.